CLINICAL TRIAL: NCT07090187
Title: Early Rehabilitation of Post Stroke Lower Limb Weakness Using Novel Assistive Device and Functional Electrical Stimulation Therapy
Brief Title: Novel Assistive Device and Functional Electrical Stimulation Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sara mohammad, Doctor Neurology specialist, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: FMASU MD106/2024
Record Dates: First submitted 2025-01-30; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-01

CONDITIONS: Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LegoPress (Active Comparator): 15 sessions of Lego Press + closed loop FES. Combined with 15 sessions of regular physiotherapy5 sessions per week, 1 per day, 3 weeks total.
  Interventions: Device: LegoPress , Novel assistive device
- Control (No Intervention): 15 sessions standard physiotherapy (regular physiotherapy): 5 sessions per week, 1 per day, 3 weeks total.

INTERVENTIONS:
Device: LegoPress , Novel assistive device — novel assistive device for rehabilitation using functional electrical stimulation
  Arms: LegoPress

SUMMARY:
Stroke causes neurological deficits, impacting walking, balance, strength, and independence, with high mortality and economic burden. Moreover, it brings serious mental and economic stress to patients and their families because of loss of independence. Current rehabilitation methods include standard therapy and electrical stimulation. This study introduces a novel hybrid approach combining use of an assistive device, the LegoPress, paired with closed-loop functional electrical stimulation for subacute stroke patients' lower limbs in a seated position, aiming to improve motor function particularly gait and balance.

DETAILED DESCRIPTION:
The LegoPress is a passive assistive device that allows patients to undergo FES therapy while remaining in seated position. This is crucial for stroke patients as in the early acute phase they are at a higher risk of falling due to balance and mobility issues. The LegoPress is equipped with potentiometers and force sensors to measure the distance and force in flexion and extension. Therefore, when the LegoPress paired with FES, it can be performed in a closed loop where a maximum current is set for patient safety and can provide flexion/extension. Then based off this current the stimulation current can be modulated according to the position desired by the clinician. It can also be an alternative to cycling FES by featuring different movement functions such as simultaneous leg press action (in tandem), gait-simulation action (closest to walking), or sequential (one leg after the other).

The efficacy of the LegoPress FES protocol has yet to be tested in the clinic and with stroke patients, this study therefore is motivated by investigating the feasibility of this proposed novel method as well as its clinical outcomes.

ELIGIBILITY:
* *Inclusion Criteria:*
* Ages 18 to 70 (max of 70 years to avoid fatigue or exhaustion in elderly patients)
* Patients with acute ischemic or hemorrhagic stroke, verified by CT or MRI
* Patients with power in the paretic lower limb synergistic extension = 2 or more on the MRC scale
* *Exclusion Criteria:*
* Patients presenting with paraplegia, ataxia, or severe sensory impairment
* Patients with subarachnoid hemorrhage
* Subjects with implanted electronic devices, such as cardiac pacemakers or any metallic implants in the lower limbs
* Patients with other severe medical comorbidities, including:
* Severe osteoarthritis
* Liver dysfunction
* Kidney dysfunction
* Cardiovascular dysfunction
* Patients with severe cognitive impairment preventing task completion, verified by a score of less than 7 on the Abbreviated Mental Test (AMT)
* Patients who are:
* Uncooperative
* Hemodynamically unstable
* Have a disturbance of consciousness
* Patients with burns or any skin lesions at the sites of stimulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy and tolerability of LegoPress device in conjunction with functional electrical stimulation (FES) on the paretic lower limb in acute stroke patients. | For each participant in intervention group: 15 sessions of Lego Press + closed loop FES. Combined with 15 sessions of regular physiotherapy5 sessions per week, 1 per day, 3 weeks total.
  Objective:
  To quantify motor function improvements and Gait performance in patients undergoing combined Lego Press + Closed-Loop FES therapy with standard physiotherapy.
  Primary Outcomes
  1. Motor Function
     Assessment Tool: Medical Research Council (MRC) scale for motor power.
  2. Gait Speed
  10-Meter Walk Test (10MWT)
  Timed Up and Go Test (TUG)
  Assessment Schedule:
  t=0: Baseline (before first session)
  t=1: Midpoint (after 7 sessions)
  t=2: Post-intervention (after 15 sessions, 3 weeks total)

SECONDARY OUTCOMES:
Over all functional improvement and Functional Independence | Each participant will undergo: 15 sessions of Lego Press + closed-loop Functional Electrical Stimulation (FES) 15 sessions of conventional physiotherapy 5 sessions/week, 1 session/day over 3 weeks
  1. Overall Motor Function
     Assessment Tool: Fugl-Meyer Assessment for Lower Extremity (FMA-LE)
     Timepoints: t=0, t=1, t=2
  2. Daily Living Functionality
     Functional Ambulation Category (FAC).
     Assessment Schedule:
     t=0: Baseline (before first session)
     t=1: Midpoint (after 7 sessions)
     t=2: Post-intervention (after 15 sessions, 3 weeks total)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Sara Mohammad Gaber Mahmoud, MD, Principal Investigator — Ainshams University
Locations (1):
- Faculty of medicine Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will be available on reasonable request near publishing